CLINICAL TRIAL: NCT00261014
Title: REcurrent VEnous Thromboembolism Risk Stratification Evaluation A Study to Develop a Clinical Prediction Rule to Predict Low Recurrence Risk in Patients With Idiopathic Venous Thromboembolism.
Brief Title: Understanding Risk Factors Involved in Developing a Second Blood Clot.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Biomerieux inc (Industry); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: 2002452-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Deep Vein Thrombosis
Keywords: Recurrent; Idiopathic; Deep Vein Thrombosis; Pulmonary Embolism; Clinical Prediction Rule; Venous Thromboembolism; Risk Factors
MeSH Terms: conditions — Venous Thrombosis; Recurrence; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a way to predict which patients diagnosed with idiopathic blood clots can safely stop warfarin therapy after six months. We will use patient characteristics, blood test results and imaging test results to identify those patients who have the lowest risk of developing a new blood clot after warfarin is stopped.

DETAILED DESCRIPTION:
The risk of recurrent VTE in patients with idiopathic VTE subsequent to three to six months of oral anticoagulant therapy remains high (5-27% per year). The risk of recurrent VTE, however, is not likely high enough to justify indefinite anticoagulation in all patients with a first idiopathic VTE due to the rate of major bleeding with oral anticoagulants (2-6% per year), the inconvenience and cost of oral anticoagulant therapy, monitoring of oral anticoagulant therapy (e.g. prescription costs, time off work to go for lab tests, parking etc) and the lifestyle limitations of oral anticoagulant therapy (avoidance of certain physical activities, dietary restrictions, avoidance of pregnancy). Further, as some have argued, perhaps all that anticoagulant therapy achieves is to delay recurrent VTE and, as a recent editorial suggested, a tailored approached is required to determine sub-groups who require lifelong anticoagulation. A means to stratify patients with idiopathic VTE to identify a group at low risk of recurrent VTE who could safely discontinue oral anticoagulants subsequent to six months of therapy would be a significant advance in the care of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Objectively proven (as previously described (8)) proximal idiopathic deep vein thrombosis or pulmonary embolism. Idiopathic will be defined as VTE occurring in the absence of fracture, plaster cast, immobilization greater than 3 days or a general anesthetic in the last three months prior to VTE diagnosis; a known deficiency of antithrombin, protein C or protein S; and malignancy in the last five years
2. Patients treated initially with a minimum of five days of heparin or low molecular weight heparin and oral anticoagulants with a target intensity of 2.0 - 3.0 with no recurrence in the subsequent six months.
3. Patients currently on oral anticoagulants

Exclusion Criteria:

1. Recurrent idiopathic VTE (i.e. ≥ 2 previous idiopathic VTE). Previous secondary VTE is not an exclusion criterion;
2. Age <18;
3. Known deficiency of proteins S, protein C or antithrombin;
4. Known, persistently positive anticardiolipin antibodies (titers > 30U/ml);
5. Known, persistently positive lupus anticoagulant;
6. Combined thrombophilic defects (e.g. homozygous for FVL or PGM, or compound heterozygous for FVL and PGM);
7. Refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with idiopathic blood clots
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2002-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adjudicated recurrent VTE during study follow-up | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD MSc, Principal Investigator — OHRI
Locations (7):
- Canada (6):
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Jewish General Hospital, Montreal, Quebec
  - Hopital du Sacre Coeur, Montreal, Quebec
- CHU de le Cavale Blanche, Brest, France

REFERENCES:
- [Derived] Wan T, Rodger M, Zeng W, Robin P, Righini M, Kovacs MJ, Tan M, Carrier M, Kahn SR, Wells PS, Anderson DR, Chagnon I, Solymoss S, Crowther M, White RH, Vickars L, Bazarjani S, Le Gal G. Residual pulmonary embolism as a predictor for recurrence after a first unprovoked episode: Results from the REVERSE cohort study. Thromb Res. 2018 Feb;162:104-109. doi: 10.1016/j.thromres.2017.11.020. Epub 2017 Dec 8. PMID 29224973
- [Derived] Rodger MA, Scarvelis D, Kahn SR, Wells PS, Anderson DA, Chagnon I, Le Gal G, Gandara E, Solymoss S, Sabri E, Kovacs J, Kovacs MJ. Long-term risk of venous thrombosis after stopping anticoagulants for a first unprovoked event: A multi-national cohort. Thromb Res. 2016 Jul;143:152-8. doi: 10.1016/j.thromres.2016.03.028. Epub 2016 Mar 29. PMID 27086275
- [Derived] Galanaud JP, Holcroft CA, Rodger MA, Kovacs MJ, Betancourt MT, Wells PS, Anderson DR, Chagnon I, Le Gal G, Solymoss S, Crowther MA, Perrier A, White RH, Vickars LM, Ramsay T, Kahn SR. Predictors of post-thrombotic syndrome in a population with a first deep vein thrombosis and no primary venous insufficiency. J Thromb Haemost. 2013 Mar;11(3):474-80. doi: 10.1111/jth.12106. PMID 23279046
- [Derived] Galanaud JP, Holcroft CA, Rodger MA, Kovacs MJ, Betancourt MT, Wells PS, Anderson DR, Chagnon I, Le Gal G, Solymoss S, Crowther MA, Perrier A, White RH, Vickars LM, Ramsay T, Kahn SR. Comparison of the Villalta post-thrombotic syndrome score in the ipsilateral vs. contralateral leg after a first unprovoked deep vein thrombosis. J Thromb Haemost. 2012 Jun;10(6):1036-42. doi: 10.1111/j.1538-7836.2012.04713.x. PMID 22646832
- [Derived] Kovacs MJ, Kahn SR, Wells PS, Anderson DA, Chagnon I, LE Gal G, Solymoss S, Crowther M, Perrier A, Ramsay T, Betancourt MT, White RH, Vickars L, Rodger MA. Patients with a first symptomatic unprovoked deep vein thrombosis are at higher risk of recurrent venous thromboembolism than patients with a first unprovoked pulmonary embolism. J Thromb Haemost. 2010 Sep;8(9):1926-32. doi: 10.1111/j.1538-7836.2010.03958.x. PMID 20561184
- [Derived] Le Gal G, Kovacs MJ, Carrier M, Do K, Kahn SR, Wells PS, Anderson DA, Chagnon I, Solymoss S, Crowther M, Righini M, Perrier A, White RH, Vickars L, Rodger M. Validation of a diagnostic approach to exclude recurrent venous thromboembolism. J Thromb Haemost. 2009 May;7(5):752-9. doi: 10.1111/j.1538-7836.2009.03324.x. Epub 2009 Feb 18. PMID 19228281
- [Derived] Rodger MA, Kahn SR, Wells PS, Anderson DA, Chagnon I, Le Gal G, Solymoss S, Crowther M, Perrier A, White R, Vickars L, Ramsay T, Betancourt MT, Kovacs MJ. Identifying unprovoked thromboembolism patients at low risk for recurrence who can discontinue anticoagulant therapy. CMAJ. 2008 Aug 26;179(5):417-26. doi: 10.1503/cmaj.080493. PMID 18725614